CLINICAL TRIAL: NCT02712242
Title: The Effects of Platelet-Rich Fibrin on Palatal Wound Healing After Free Gingival Graft Harvesting: A Comparative Randomized Controlled Clinical Trial
Brief Title: PRF for Accelerating Palatal Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Onur Ozcelik, Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CukurovaU8
Record Dates: First submitted 2016-03-09; First posted 2016-03-18 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Platelet Rich Fibrin (Experimental): PRF was laid directly on the palatal wound immediately after harvesting the tissue graft and stabilized
  Interventions: Other: Platelet Rich Fibrin
- Butyl cyanoacrylate (Active Comparator): Butyl cyanoacrylate was directly applied on the palatal wound after harvesting the tissue graft
  Interventions: Other: Butyl cyanoacrylate
- Wet Gauze (Placebo Comparator): Wet Gauze was placed for 1 minute on the palatal wound after harvesting the tissue graft
  Interventions: Other: Wet gauze

INTERVENTIONS:
Other: Platelet Rich Fibrin — Immediate and delayed bleeding, pain, epithelialization, feeding habits and sensation scores were recorded after PRF placing on palatal wounds.
  Arms: Platelet Rich Fibrin
Other: Butyl cyanoacrylate — Immediate and delayed bleeding, pain, epithelialization, feeding habits and sensation scores were recorded after Butyl Cyanoacrylate application on palatal wounds.
  Arms: Butyl cyanoacrylate
Other: Wet gauze — Immediate and delayed bleeding, pain, epithelialization, feeding habits and sensation scores were recorded after wet gauze pressure on palatal wounds.
  Arms: Wet Gauze

SUMMARY:
Backgroung: Various agents are used to reduce post-operative complications associated with palatal donor site surgery for free gingival graft (FGG) harvesting. This study was conducted to evaluate the effects of platelet-rich fibrin (PRF) on palatal wound healing.

DETAILED DESCRIPTION:
125 patients with isolated recessions were treated. The connective tissue graft was obtained by the de-epithelialization of a free gingival graft in both groups. Three different hemostatic treatments were randomized; PRF with cyanoacrilate adhesive (PRF group, n:42), cyanoacrilate adhesive alone (BC group, n:42) and sterile wet gauze compression (WG group, n:41). Immediate and delayed bleeding, pain, epithelialization, feeding habits and sensation scores were recorded for different time points.

ELIGIBILITY:
Inclusion Criteria:

* no contraindications for periodontal surgery;
* full-mouth plaque score of <10%
* full-mouth bleeding score of <15%.

Exclusion Criteria:

* previously undergone surgery for a graft harvested from the palate
* presence of systemic disease or taking medication known to interfere with periodontal health
* smokers
* possible coagulation disorders

Ages: 21 Years to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2013-11; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Epithelialization | One month
  Assessed according to the toluedine blue coloring

SECONDARY OUTCOMES:
Sensibility disorders | One month
  visual analogue scale scores
feeding habits | One month
  visual analogue scale scores
Delayed bleeding | 1 week
  Bleeding assesment for post-operative one week
Immediate Bleeding | 1 hour
  Bleeding assesment for post-operative one hour
Pain | 3 months
  Visual Analague Scale scores

CONTACTS AND LOCATIONS:
Overall Officials: Onur Ozcelik, Ph D, Study Director — Cukurova University, Professor

IPD SHARING:
Plan to Share IPD: No